CLINICAL TRIAL: NCT04079647
Title: Immune Checkpoint Inhibitor Therapy- Induced Endocrinopathy and Metabolic Diseases -a Case Series of Taiwanese Patients
Brief Title: Immune Checkpoint Inhibitor Therapy- Induced Endocrinopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805155RIND
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Endocrinopathy
MeSH Terms: conditions — Endocrine System Diseases | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with endocrinopathy after immunotherapy: Patient with endocrinopathy after immunotherapy
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — Patients receive immunotherapy for cancer treatment
  Other Names: Immune blockade therapy

SUMMARY:
To review cases from NTUH who developed endocrinopathy and metabolic diseases after immunotherapy, and statistically analyzed their age, clinical presentation, image findings, treatment and its response.

DETAILED DESCRIPTION:
Immune checkpoint blockade-based immunotherapy is a new modality of cancer treatment with a unique mechanism that has gained increased numbers of indication and is now used in several cancer types. However, immune-related adverse events (irAEs) emerge as a new entity of diseases involving one or multiple organ systems. irAEs could result in interruption of immunotherapy, morbidities of patients or even death. Among various manifestations of irAEs, endocrinopathy and metabolic diseases are rare but important, and require prompt diagnosis and treatment to avoid life-threatening conditions.

Thus, we intend to review cases from NTUH who developed endocrinopathy and metabolic diseases after immunotherapy, and statistically analyzed their age, clinical presentation, image findings, treatment and its response. We will also review literatures to evaluate the difference and similarity from previous diagnostic and treatment experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive immunotherapy in NTUH and develop endocrinopathy after therapy

Exclusion Criteria:

* Patients less than 20 years old. Patients who are pregnant

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive immunotherapy in NTUH and develop endocrinopathy after therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-03 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes of endocrine profiles | 10 year
  Changes of serum fT4 TSH Glucose A1C ACTH cortisol LH FSH estradiol progesterone GH IGF1 prolactin

SECONDARY OUTCOMES:
Treatment response of the cancer after immunotherapy | 10 years
  The changes of size and extent of the tumors

CONTACTS AND LOCATIONS:
Overall Officials: Shyang-Rong Shih, MD, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- Shyang-Rong Shih, Taipei, Taiwan